CLINICAL TRIAL: NCT07155070
Title: Kera Sol Post-LASIK: A Benefit Study
Brief Title: Efficacy of Kera Sol Tears on Signs and Symptoms of Surgical Temporary Ocular Discomfort Syndrome (STODS) in Subjects Following LASIK
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Vance Thompson Vision (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Surface IIT
Record Dates: First submitted 2025-08-26; First posted 2025-09-04 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Intervention Model Description: Two-arm randomized study evaluating the impact of, Kera Sol tears on the signs and symptoms of STODS in 60 patients who underwent bilateral LASIK. Both groups will be prescribed the standard of care post-operative prescription combination steroid and antibiotic drop.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Kera Sol (Active Comparator): Subjects will be randomized to administer the study drop (Kera Sol) dosed QID for 14 days.
  Interventions: Drug: Kera Sol Eye Drops
- Standard of Care (No Intervention): No Kera Sol drops

INTERVENTIONS:
Drug: Kera Sol Eye Drops — Eye drops
  Arms: Kera Sol

SUMMARY:
Collecting data using Kera Sol tear usage during the initial two-week post-operative period after Laser-Assisted In Situ Keratomileusis (LASIK) has on the signs and symptoms of surgical temporary ocular discomfort syndrome (STODS)

DETAILED DESCRIPTION:
Prospective, single-site, two-arm randomized study evaluating the impact of, Kera Sol tears on the signs and symptoms of STODS in 60 patients who underwent bilateral LASIK. Both groups will be prescribed the standard of care post-operative prescription combination steroid and antibiotic drop. Additionally, subjects will be randomized to administer the study drop (Kera Sol) dosed QID for 14 days.

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to sign the informed consent form (ICF)
* Be at least 18 years of age at the screening visit
* Be undergoing LASIK treatment in both eyes
* Be literate and able to complete questionnaires independently
* Be able and willing to use the study drug and participate in all study assessments and visits
* Have provided verbal and written informed consent

Exclusion Criteria:

* Use of topical prescription dry eye medications such as lifitegrast, cyclosporine, loltilaner, etc.
* Have a break in the integrity of the corneal epithelium such as a persistent corneal epithelial defect, or corneal ulcer.
* Have presence of corneal pathology that may interfere with LASIK outcomes
* Active infectious, ocular or systemic disease
* Have a history of ocular inflammation or macular edema
* Have had clinically significant active infectious keratitis in the past 3 months 7. -Have history of prior refractive surgery
* Have placement of temporary punctal plugs in the past 1 month or current presence of permanent punctal plugs at time of screening
* Patients with usual relative and absolute contraindications for LASIK surgery (Patients with severe dry eye, recurrent corneal erosion, uncontrolled Glaucoma, collagen vascular disorders, keratoconus or signs of keratoconus, uncontrolled Diabetes, Herpes)
* Autoimmune or immunodeficiency diseases
* Pregnant or nursing women
* Patients with history of previous ocular surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Change in Baseline of Corneal Staining | 14 days
  Using the National Eye Institute (NEI) scale system. The NEI scale system for grading fluorescein staining divides the corneal and conjunctival surfaces. The conjunctival surface is divided into 6 areas and the corneal surface is divided into 5 areas. A standardized grading system of 0 to 3 is used for each of areas on cornea and conjunctiva.
  The maximum staining score for the cornea is 15, and for conjunctiva, the maximum score is 18. The values above 3 is considered abnormal for cornea or conjunctiva in each eye. Grade 0 (i.e., no staining) indicates normal cornea or normal conjunctiva
  Grade 3 (i.e., highest severity staining) indicates severe ocular surface damage
  NEI Scale ranges from 0-4. Grade 0 = no dots; Grade 1 = 1-15 dots; Grade 2 = 16-30 dots, and Grade 3 = 31 or > dots.

CONTACTS AND LOCATIONS:
Overall Officials: Dan Terveen, MD, Principal Investigator — Vance Thompson Vision Clinic Prof. LLC
Locations (1):
- Vance Thompson Vision Clinic, Prof. LLC, Sioux Falls, South Dakota, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF

DOCUMENTS (2):
  • Study Protocol (2025-04-10): https://cdn.clinicaltrials.gov/large-docs/70/NCT07155070/Prot_000.pdf
  • Informed Consent Form (2025-06-26): https://cdn.clinicaltrials.gov/large-docs/70/NCT07155070/ICF_001.pdf